CLINICAL TRIAL: NCT00512577
Title: Transfusion Alternatives Pre-operatively in Sickle Cell Disease
Brief Title: Transfusion Alternatives Pre-operatively in Sickle Cell Disease (TAPS)
Acronym: TAPS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated by Trial Steering Committee.
Sponsor: NHS Blood and Transplant (Other Government)
Collaborators: British Medical Research Council (Other Government); University of York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BS02/4/RB31; ISRCTN:00862331
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; pre-operative transfusion; blood transfusion
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Patients will not receive a pre-operative transfusion.
  Interventions: Other: Red blood cell transfusion
- B (Active Comparator): Patients will receive a pre-operative blood transfusion. Those presenting with an admission Hb of less than 9g/dL will receive a simple (also called a 'top-up') transfusion, those presenting with an admission Hb of more than or equal to 9g/dL will undergo a partial exchange transfusion.
  Interventions: Other: Red blood cell transfusion

INTERVENTIONS:
Other: Red blood cell transfusion — Pre-operative red blood cell transfusion

SUMMARY:
TAPS is a sequential trial which aims to investigate whether the administration of a blood transfusion pre-operatively to patients with sickle cell disease (HB SS or Hb SB0 thal)having low or medium risk elective surgery increases or decreases the overall rate of peri-operative complications. The proportion of patients with peri-operative complications in two randomised groups of transfused and untransfused patients will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease, either Hb SS or Hb SB0 thal, confirmed by Hb electrophoresis, Deoxyribonucleic Acid (DNA) analysis or High Performance Liquid Chromatography (HPLC)
* At least 24 hourse and no more than 14 days before surgery and a date for surgery has been given
* Surgery to be low or medium risk
* Surgery to be with general or regional anaesthesia
* Written informed consent from patient/parent/guardian is given
* More than six months since previous TAPS trial surgery.

Exclusion Criteria:

* Having a procedure involving intravascular contrast radiography or an imaging procedure
* On a regular blood transfusion regime
* Had a blood transfusion within the last three months
* The planned procedure involves local anaesthetic only
* Haemoglobin level at randomisation less than 6.5g/dL
* Children with a clinical history of stroke (history of silent infarcts would not preclude randomisation)
* Acute chest syndrome within the last six months, or patient has ever required intubation and mechanical ventilation for treatment of acute chest syndrome
* Oxygen saturation at randomisation less than 90%
* Patient is on renal dialysis
* Already entered twice into the TAPS trial
* The physician is unwilling to randomise the patient (such patients will be entered into a trial log).

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The frequency of all clinically significant complications in sickle Cell patients (Hb SS or SB0 thal) undergoing low or medium risk planned surgery. | Between randomisation and 30 days post surgery, inclusive.

SECONDARY OUTCOMES:
1. Complications included in the primary outcome, plus red cell alloimmunisation. | Up to 3 months post surgery.
2. Total days in hospital, to include hours/days spent having pre-operative transfusion, days on intensive care and high dependency units, and other wards. | Up to 30 days post surgery, inclusive.
3. Re-admission or failure to discharge. | Up to 30 days post surgery.
Number of red cell units received. | Intra and post-operatively.
Health economic analysis: differential health service costs of routine transfusion relative to control, plus quality adjusted survival and treatment cost-effectiveness and benefits in QOL years. | Up to 30 days post surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna M Williamson, MRCP,MRCPath, Study Chair — University of Cambridge and NHSBT; Sally C Davies, MRCP,MRCPath, Study Chair — Imperial College, University of London and Central Middlesex Hospital
Locations (1):
- NBS/MRC Clinical Studies Unit, National Blood Service, Cambridge, Cambridgeshire, United Kingdom